CLINICAL TRIAL: NCT06733662
Title: The Effect of Motivational Interviewing-Based Education on Treatment Adherence and Self-Care Agency in COPD Patients: A Randomized Controlled Trial
Brief Title: The Effect of Motivational Interviewing-Based Education on Treatment Adherence and Self-Care Agency in COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaraş İstiklal University (Other)
Responsible Party: Principal Investigator, Yasemin Sazak, Assistant Professor, Kahramanmaraş İstiklal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstiklalU-YSazak-003
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Motivational Interviewing; COPD
Keywords: Self-care; Treatment adherence; Education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education-based motivational interviewing Group (Experimental): Patients in the intervention group will be given COPD education lasting approximately 45-50 minutes in a single session in line with the education booklet and by evaluating the pre-test data. On the 3rd day, the first session of motivational interview will be held. On the 5th day and 7th day and 15th day, motivational interview sessions will continue with the patients.
  Interventions: Behavioral: Experimental: Education-based motivational interviewing Group
- Control group (No Intervention): There will be no intervention for individuals in this group.

INTERVENTIONS:
Behavioral: Experimental: Education-based motivational interviewing Group — The Effect of Motivational Interviewing-Based Education on Treatment Adherence and Self-Care Agency in COPD Patients
  Arms: Education-based motivational interviewing Group

SUMMARY:
This randomized controlled trial will be conducted to evaluate the effect of education and motivational interviewing on treatment adherence and self-care power in COPD patients.

Hypotheses of the Study; H1: Education and motivational interviewing in COPD patients increase treatment adherence in patients.

H2: Education and motivational interviewing in COPD patients increase self-care power in patients.

There will be two groups in the study: control and intervention groups. Before the intervention, pre-test data will be collected in the control and intervention groups. After the intervention, post-test data will be collected in both groups in line with the data collection forms.

DETAILED DESCRIPTION:
In line with the randomization list, patients will be assigned to the intervention and control groups in line with the inclusion criteria. Pre-test data will be collected face-to-face in the intervention group in accordance with the data collection forms. After collecting the pre-test data, the patient will be allowed to rest for about 10 minutes, and then COPD training will be given to the patient in a single session lasting about 45-50 minutes in line with the training booklet and by evaluating the pre-test data. The education booklet will be given to the patient. On the 3rd day, the first session of motivational interview will be held. On the 5th day and 7th day and 15th day, motivational interview sessions will continue with the patients. During the motivational interview, patients will be supported in line with the training booklet. On the 30th day, the patient will be interviewed face-to-face and post-test data will be collected.

Patients in the control group will be interviewed and no intervention will be made after the pre-tests are applied. Patients in the control group will continue their routine controls. In the final test (1st month), an appointment date will be set with the patient and the final test data will be collected face-to-face.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COPD for at least 6 months
* Admitted to the chest clinic
* No communication problems
* Patients who volunteered to participate in the study.

Exclusion Criteria:

* In the period of exacerbation
* Uncooperative due to dyspnea
* With a malignant disease
* Patients with a confirmed diagnosis of psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Morisky 8-item Medication Adherence Scale | 0 days
  It is a scale that assesses self-reported medication use behaviors of the patient. It consists of eight questions. A validation study in Turkish was conducted by Oğuzülgen et al. in 2014. While the first seven questions are answered as "yes/no", the eighth question is answered on a five-point Likert scale as "never/rarely", "sometimes", "sometimes", "usually" and "always". Morisky 8-item medication adherence scale is calculated between 0-8 points.
Morisky 8-item Medication Adherence Scale | 30 days
  It is a scale that assesses self-reported medication use behaviors of the patient. It consists of eight questions. A validation study in Turkish was conducted by Oğuzülgen et al. in 2014. While the first seven questions are answered as "yes/no", the eighth question is answered on a five-point Likert scale as "never/rarely", "sometimes", "sometimes", "usually" and "always". Morisky 8-item medication adherence scale is calculated between 0-8 points.
Self-care Agency Scale | 0 days
  The scale was developed by Kearney and Fleischer and its validity and reliability study in Turkey was conducted by Nahcivan in 1993. In Nahcivan's study, the Cronbach's alpha coefficient of the scale was found to be 0.92. This scale, in which individuals self-assess their ability or power to perform self-care actions, consists of 35 items. The maximum score to be obtained from the scale is 140. As the score obtained from the scale increases, the self-care power of the patients also increases.
Self-care Agency Scale | 30 days
  The scale was developed by Kearney and Fleischer and its validity and reliability study in Turkey was conducted by Nahcivan in 1993. In Nahcivan's study, the Cronbach's alpha coefficient of the scale was found to be 0.92. This scale, in which individuals self-assess their ability or power to perform self-care actions, consists of 35 items. The maximum score to be obtained from the scale is 140. As the score obtained from the scale increases, the self-care power of the patients also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Istiklal Universty, Kahramanmaraş, Turkey (Türkiye)